CLINICAL TRIAL: NCT01414374
Title: Prevalence of Genetic Polymorphisms of DMT1 and Ferroportin Enzymes in Adults With Anemia by Iron Deficiency, and Its Influence on the Efficacy of Conventional and Herbal Treatments
Brief Title: Hibiscus Sabdariffa and Centella Asiatica in the Treatment of Anemia by Iron Deficiency
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Casa Espirita Terra de Ismael (Other)
Collaborators: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Fabio Carmona, Assistant Professor, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ANEMIA2011
Record Dates: First submitted 2011-08-09; First posted 2011-08-11 (Estimated); Last update posted 2015-02-13 (Estimated); Status verified 2015-02

CONDITIONS: Iron Deficiency Anemia
Keywords: iron; anemia; herbal medicine; phytotherapy; Centella asiatica; Hibiscus sabdariffa
MeSH Terms: conditions — Anemia, Iron-Deficiency; Anemia | interventions — Phytotherapy; Iron

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Iron (Active Comparator)
  Interventions: Drug: Iron
- Herbal (Experimental)
  Interventions: Drug: Herbal medicine

INTERVENTIONS:
Drug: Herbal medicine — Patients will receive a combination of Hibiscus sabdariffa (powdered dry plant), 200 mg, BID, and Centella asiatica tincture, 40 drops, BID, for 6 weeks.
  Arms: Herbal
Drug: Iron — Patients will receive iron sulphate, 500 mg, BID, plus orange juice, for 6 weeks.
  Arms: Iron

SUMMARY:
The study aims to investigate the prevalence of genetic polymorphisms in adults with iron deficiency and anemia, and the responses to two different treatments: iron sulphate and a composite herbal medicine (Hibiscus sabdariffa plus Centella asiatica). The main outcome will be hemoglobin, measured before and after 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 y and < 50 y
* A diagnostic of iron deficient anemia

Exclusion Criteria:

* Severe anemia
* Treatment interruption for more than 25% of the 6 weeks
* New onset severe adverse symptoms or events
* Patient's request

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2012-01; Primary Completion 2012-12 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Hemoglobin | 6 weeks
  Hemoglobin will be measured before treatment and after 6 weeks of treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Laboratorio M. F. Teixeira, Monte Santo de Minas, Minas Gerais, Brazil